CLINICAL TRIAL: NCT01875380
Title: A Phase II Study of Single-agent Regorafenib in the First Line Treatment of Frail and/or Unfit for Polychemotherapy Patients With Metastatic Colorectal Cancer (mCRC)
Brief Title: Regorafenib in Frail and/or Unfit for Chemotherapy Patients With Metastatic Colorectal Cancer
Acronym: REFRAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-13-01; 2013-000236-94 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Neoplasms; Metastatic Disease
Keywords: metastatic colorectal cancer; frail and unfit patient; regorafenib
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib (Experimental): Regorafenib will be administered orally at the initial dosage of 160 mg per day for 3 weeks,followed by one week of rest, according to the 3/1 regimen.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib

SUMMARY:
The purpose of this study is to assess the efficacy and safety of single-agent regorafenib in the first line treatment of frail and/or unfit for polychemotherapy patients with metastatic colorectal cancer (mCRC)

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the informed consent form.
2. The patient must be able to understand the information and state expressly his or her desire to take part in the study.
3. Age > 18 years.
4. Patients with histologically or cytologically documented adenocarcinoma of the colon or rectum who have not been previously treated systemically for advanced disease. Patients can have received fluoropyrimidine-based adjuvant therapy if the last dose was taken at least 6 months prior to study entry.
5. Patients who are frail and/or unfit for polychemotherapy owing to the presence of one or more of the following criteria:

   1. Patients with dependence in activities of daily living owing to the presence of comorbidities other than those resulting from the deterioration caused by the neoplastic disease.
   2. Presence in the patient's medical history of three or more of the following comorbidities, even if they are under control with proper treatment:

      * Congestive heart failure
      * Other chronic cardiovascular diseases
      * Chronic obstructive pulmonary disease
      * Cerebrovascular disease
      * Peripheral neuropathy
      * Chronic kidney failure
      * Hypertension
      * Diabetes mellitus
      * Systemic vasculitis
      * Severe arthritis
   3. Presence of geriatric syndromes such as age > 85 years, faecal or urinary incontinence, spontaneous bone fractures, mild and moderate dementia, or patients who fall repeatedly.
6. Existence of at least one measurable unidimensional lesion using CT or MRI based on the Response Evaluation Criteria in Solid Tumors criteria (RECIST), version 1.1
7. Overall Eastern Cooperative Oncology Group (ECOG) performance less than or equal to 2
8. Patient's commitment to compliance with the oral medication throughout the duration of the study
9. Life expectancy of at least 3 months
10. Adequate bone marrow, renal and hepatic function, defined as:

    1. Neutrophils > 1500/mm3
    2. Platelets > 100,000/mm3
    3. Creatinine clearance > 30 ml/min
    4. Hemoglobin ≥ 9 gr/dl
    5. Bilirubin levels < 2.5 x ULN
    6. Aspartate aminotransferase (AST) and alanine transaminase (ALT) levels < 3 x ULN (if liver metastases < 5 x ULN)

Exclusion Criteria:

1. Prior treatment with regorafenib.
2. Assignment prior to treatment during this study. Patients who are permanently withdrawn from participation in the study treatment will not be allowed to return to it.
3. Prior or concurrent presence of another neoplastic disease that is different in terms of tumour site and histology of the colorectal cancer in the 5 years prior to the inclusion of the patient in the study, except in situ cervical cancer, superficial bladder carcinoma [Ta (non-invasive), Tis (carcinoma in situ) and T1 (tumour invades lamina propria)] and non-melanoma skin tumours.
4. Presence or history of brain metastases or meningeal tumours.
5. Major surgery, open biopsy or traumatic injury within 28 days prior to the start of patient treatment with the study medication.
6. Extended-field radiotherapy within 4 weeks prior to randomisation or limited-field radiotherapy in the previous 2 weeks. Patients must have recovered from all treatment-related toxicities.
7. Pregnant or breastfeeding women. Women of childbearing age must use adequate contraception. Women of childbearing age must have a negative pregnancy test within 7 days prior to starting with the study medication.
8. Women of childbearing age and men who wish to take part in the study must agree to use adequate contraception from the signing of the informed consent until at least 3 months after stopping the study medication. The investigator or the person designated by him or her will ensure and advise as to the contraceptive methods that should be used. Appropriate contraceptive methods include abstinence, oral contraceptives, transdermal patches and injections of sustained-release progestin (starting at least 4 weeks before administration of the IMP), double-barrier method: condom or female condom (diaphragm or cervical/vaginal condom) plus spermicide, intrauterine device (IUD), intrauterine system, implant or vaginal ring (in place at least 4 weeks before administration of the IMP) or male partner sterilization (vasectomy with documentation of azoospermia) prior to inclusion of the woman in the trial if he is the woman's only sexual partner.
9. Active congestive heart failure class 2 or higher on the New York Heart Association (NYHA) scale.
10. Unstable angina (angina symptoms at rest), new-onset angina (having appeared in the past 3 months) or acute myocardial infarction that has occurred in the 6 months prior to starting with the study medication.
11. Cardiac arrhythmias that require anti-arrhythmic therapy (only beta blockers and digoxin would be allowed as concomitant medication for these patients).
12. Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg) despite proper medical management.
13. Patients with phaeochromocytoma.
14. Pleural effusion or ascites that cause breathing difficulties (dyspnoea of grade ≥2 of the CTC).
15. Accidents (including transient ischaemic attacks), deep vein thrombosis or pulmonary thromboembolism that have occurred in the 6 months prior to starting with the study medication.
16. Active infection > grade 2 based on the NCI CTC, v. 4.0.
17. Human immunodeficiency virus (HIV) infection.
18. Active hepatitis B or C, or hepatitis B or C infection that requires treatment with antiviral drugs.
19. Patients with severe mental disorders that require medication.
20. Presence or history of brain metastases or meningeal tumours.
21. History of organ transplants.
22. Patients with evidence or history of bleeding diathesis. Any bleeding or bleeding event > Common Toxicity Criteria for Adverse Effects (CTCAE) grade 3 in the 4 weeks prior to starting with the study medication.
23. Presence of unhealed wounds, ulcers or bone fractures.
24. Kidney failure requiring haemodialysis or peritoneal dialysis.
25. Dehydration based on NCI CTC criteria, version 4, of > 1.
26. Substance abuse or a history of medical, social or psychological conditions that may interfere with study participation or compliance with the efficacy and safety assessments planned in the study.
27. Known hypersensitivity to regorafenib or any of its excipients.
28. Presence of any disease or medical condition that might interfere with patient safety or may compromise treatment compliance with it.
29. Interstitial lung disease with signs and symptoms present at the time of signing the informed consent.
30. Patients who are unable to swallow oral medication.
31. Persistent proteinuria > grade 3 based on the NCI CTC, version 4.0 (> 3.5 g/24 hours).
32. Intestinal malabsorption syndrome.
33. Close personal relationship with the research staff, such as family members of the investigator or dependents (e.g. employees or students of the research centre).
34. Unresolved toxicity grade > 1 based on the NCI CTC, version 4.0 (except alopecia), related to any previous therapy or procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months | 6 months

SECONDARY OUTCOMES:
Objective response rate | 30 months
Disease control rate | 30 months
Time to response | 30 months
Time to progression | 30 months
Progression-free survival | 30 months
Time to treatment failure | 30 months
Response duration | 30 months
Duration of stable disease | 30 months
Overall survival | 30 months
Incidence and severity of Adverse Events (NCI CTC, version 4.0) | 30 months
Changes in laboratory values (transaminases, bilirubin, lactate dehydrogenase (LDH), anaemia,neutropenia and thrombocytopenia) | 30 months
Change in vital signs (weight loss and hypertension) | 30 months
Incidence of dose adjustments and compliance | 30 months
Incidence of concomitant medication | 30 months
Changes in ECOG performance status over time from baseline | 30 months

OTHER OUTCOMES:
microRNA expression levels and their correlation with tumour-efficacy parameters (objective response rate, progression-free survival and overall survival), as well as toxicity | 30 months
Biomarkers associated with cell and tumour growth and/or the mechanism of action of regorafenib and their correlation with patients' clinical progression for efficacy and safety parameters. | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Carrato, MD-PhD, Study Chair — Ramon y Cajal University Hospital; Enrique Grande, MD, Study Chair — Ramon y Cajal University Hospital
Locations (1):
- Spanish Cooperative Group for Digestive Tumour Therapy (TTD), Madrid, Spain

REFERENCES:
- See also: Related Info — http://www.ttdgroup.org